CLINICAL TRIAL: NCT03491878
Title: Three Dimension Laparoscopic Versus Open Surgery for Gallbladder Carcinoma. A Randomized Clinical Trial
Brief Title: Three Dimension Laparoscopic Versus Open Surgery for Gallbladder Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Renyi Qin, Professor, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TJDBPS05
Record Dates: First submitted 2018-04-01; First posted 2018-04-09 (Actual); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Gallbladder Cancer; Surgery
MeSH Terms: conditions — Gallbladder Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D approach (Experimental): Three dimensional laparoscopic cholecystectomy including segments IVB and V
  Interventions: Procedure: Three dimensional laparoscopic
- open approach (Active Comparator): Open cholecystectomy including segments IVB and V
  Interventions: Procedure: Open

INTERVENTIONS:
Procedure: Three dimensional laparoscopic — Three dimensional laparoscopic cholecystectomy including segments IVB and V
  Arms: 3D approach
Procedure: Open — Open cholecystectomy including segments IVB and V
  Arms: open approach

SUMMARY:
Introduction: Surgery is the only potential curative approach for the highly lethal gallbladder carcinoma. The laparoscopic surgery has developed rapidly since invented. As a kind of minimally invasive surgery, laparoscopic cholecystectomy including segmentg IVB and V is preferred by most of surgeons. There have been studies comparing intraoperative blood loss, postoperative morbidity, length of hospital stay and costs of laparoscopic cholecystectomy over open surgery. However, randomized controlled trials are still lacking but clearly required to reveal whether the laparoscopic approach or the open surgery is the better option for treating gallbladder carcinoma. We hypothesize that incidence of postoperative complications is lower, and time to functional recovery is shorter after laparosopic compared with open approach, even in an enhanced recovery setting.

Methods/design: We designed this prospective, randomized, controlled trial with two treatment approaches, laparoscopic versus open surgery for gallbladder carcinoma. The trial hypothesis is that laparoscopic approach has advantages in postoperative recoveries and be equivalent in operation time, oncological results and long-term follow-up compared with open counterpart. The duration of the entire trial is four years including prearrangement, follow-up and analyses.

Discussion: Although several studies have discussed different surgical approaches for gallbladder carcinoma treatment, this trial will be a thorough RCT comparing laparoscopic and open surgery for gallbladder carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven gallbladder carcinoma.
2. Highly presumed malignancy with difficulties to obtain histological evidence.
3. Preoperative staging work up performed by upper abdomen enhanced CT scan and showed no vessel involvment.
4. The subject understands the nature of this trial and willing to comply.
5. Ability to provide written informed consent.
6. Patients treated with curative intent in accordance to international guidelines.

Exclusion Criteria:

1. Distant metastases: peritoneal carcinomatosis, liver metastases, distant lymph node metastases, involvement of other organs.
2. Patients with high operative risk as defined by the American Society of Anesthesiologists (ASA) score >4.
3. Synchronous malignancy in other organs.
4. Palliative surgery.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-05-01 (Estimated); Primary Completion 2021-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Operation time | 24 months
  Operation time is definied as the from either skin incision or trocar placement to the entire skin closure.
Estimated blood loss | 24 months
  EBL is defined as the blood loss during the surgical procedure
Intraoperative blood transfusion | 24 months
  IBT is defined as whether the subjects receive blood transfusion during the surgical procedure
Length of stay | 24 months
  LOS is defined as the days between the surgery and hospital discharged
Complication rate | 24 months
  Complication rate is defined as the number of subjects developed complication divided the total subjects number
R0 rescetion rate | 24 months
  R0 rescetion rate for the carcinoma

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided